CLINICAL TRIAL: NCT02116530
Title: Olanzapine for the Prevention of Chemotherapy Induced Nausea and Vomiting (CINV) in Patients Receiving Highly Emetogenic Chemotherapy (HEC): A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Antiemetic Therapy With or Without Olanzapine in Preventing Chemotherapy-Induced Nausea and Vomiting in Patients With Cancer Receiving Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A221301; NCI-2014-00446 (Other: NCI Clinical Trial Reporting Program); U10CA031946 (NIH)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic/Lymphoid Cancer; Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Hematologic Neoplasms; Nausea; Vomiting | interventions — Olanzapine; Drug Therapy; Cisplatin; Cyclophosphamide; Doxorubicin; Ondansetron; Granisetron; Palonosetron; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine + Chemotherapy + Antiemetic treatment (Experimental): Patients will receive the chemotherapy drugs cisplatin or cyclophosphamide and doxorubicin as well as the following anti-nausea/vomiting drugs:
  * Ondansetron (8 mg orally or intravenously) or granisetron (1 mg intravenously or 2 mg orally) or palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (12 mg orally on the day of chemotherapy and 8 mg orally days 2, 3, 4 post chemotherapy), plus
  * Fosaprepitant (150 mg intravenously on the day of chemotherapy) or aprepitant (125 mg orally on the day of chemotherapy and 80 mg orally on days 2 and 3 post chemotherapy), plus
  * olanzapine (10 mg orally on the day of chemotherapy and 10 mg orally on days 2, 3, 4 post chemotherapy)
  Interventions: Drug: Olanzapine; Drug: Chemotherapy (cisplatin or cyclophosphamide and doxorubicin); Drug: Antiemetic treatment (ondansetron or granisetron or palonosetron; plus dexamethasone; plus fosaprepitant or aprepitant)
- Placebo + Chemotherapy + Antiemetic treatment (Active Comparator): Patients will receive the chemotherapy drugs cisplatin or cyclophosphamide and doxorubicin as well as usual anti-nausea/vomiting drugs:
  * Ondansetron (8 mg orally or intravenously) or granisetron (1 mg intravenously or 2 mg orally) or palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (12 mg orally on the day of chemotherapy and 8 mg orally days 2, 3, 4 post chemotherapy), plus
  * Fosaprepitant (150 mg intravenously on the day of chemotherapy) or aprepitant (125 mg orally on the day of chemotherapy and 80 mg orally on days 2 and 3 post chemotherapy), plus
  * placebo
  Interventions: Drug: Chemotherapy (cisplatin or cyclophosphamide and doxorubicin); Drug: Antiemetic treatment (ondansetron or granisetron or palonosetron; plus dexamethasone; plus fosaprepitant or aprepitant); Other: Placebo

INTERVENTIONS:
Drug: Olanzapine — oral
  Arms: Olanzapine + Chemotherapy + Antiemetic treatment
Drug: Chemotherapy (cisplatin or cyclophosphamide and doxorubicin) — oral or IV
Drug: Antiemetic treatment (ondansetron or granisetron or palonosetron; plus dexamethasone; plus fosaprepitant or aprepitant) — oral or IV
Other: Placebo — oral
  Arms: Placebo + Chemotherapy + Antiemetic treatment

SUMMARY:
This randomized phase III trial studies antiemetic therapy with olanzapine to see how well they work compared to antiemetic therapy alone in preventing chemotherapy-induced nausea and vomiting in patients with cancer receiving highly emetogenic (causes vomiting) chemotherapy. Antiemetic drugs, such as palonosetron hydrochloride, ondansetron, and granisetron hydrochloride, may help lessen or prevent nausea and vomiting in patients treated with chemotherapy. Olanzapine may help prevent chemotherapy-induced nausea and vomiting by blocking brain receptors that appear to be involved in nausea and vomiting.

DETAILED DESCRIPTION:
Patients with cancer may receive chemotherapy that may cause nausea and vomiting. The purpose of this study is to determine if the use of olanzapine in combination with antiemetic therapy can significantly reduce nausea and vomiting in a large number of patients receiving chemotherapy. Patients are randomized to one of two treatment arms. Please see the "Arms and Intervention" sections for more detailed information. The primary objective is to compare the number of patients with no nausea for the acute (0-24 hours post-chemotherapy), delayed (24-120 hours post-chemotherapy) and overall periods (0-120 hours post-chemotherapy) for patients receiving HEC. The secondary objectives are:

1. To compare the complete response (CR) (no emetic episodes and no use of rescue medication) in the acute, delayed and overall periods
2. To compare the incidences of potential toxicities ascribed to olanzapine

Protocol treatment is to begin ≤ 14 days of registration. Patients will receive treatment on Days 1-4. Patients will be permitted to take rescue therapy of the treating investigator's choice for nausea and/or emesis/retching, based on clinical circumstances. After completing treatment, patients will be monitored for side effects.

ELIGIBILITY:
* Diagnosis of malignant disease
* No prior chemotherapy and scheduled to receive HEC (either cisplatin-containing regimen or anthracycline + cyclophosphamide [AC])

  * Cisplatin at a dose of ≥70mg/m^2, with or without other chemotherapy agent(s) OR
  * Anthracycline (60 mg/m^2) plus cyclophosphamide(600 mg/m^2)
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Required Initial Laboratory Values ≤ 120 days prior to registration

  * Serum Creatinine ≤2.0 mg/dL
  * Serum glutamic oxaloacetic transaminase (SGOT) or Serum glutamic oxaloacetic transaminase (SGPT) ≤3 x Upper Limit of Normal (ULN)
  * Absolute neutrophil count (ANC) ≥1500/mm^3
* No nausea or vomiting ≤ 24 hours prior to registration
* Negative pregnancy test (serum or urine) done ≤7 days prior to registration, for women of childbearing potential only (per clinician discretion)
* No severe cognitive compromise
* No known history of CNS disease (e.g. brain metastases, seizure disorder)
* No treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, phenothiazine or butyrophenone ≤30 days prior to registration or planned during protocol therapy
* No chronic phenothiazine administration as an antipsychotic agent (patients may receive prochlorperazine and other phenothiazines as rescue anti-emetic therapy)
* No concurrent use of amifostine
* No concurrent abdominal radiotherapy
* No concurrent use of quinolone antibiotic therapy
* No chronic alcoholism (as determined by the investigator)
* No known hypersensitivity to olanzapine
* No known cardiac arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within the previous six months.
* No history of uncontrolled diabetes mellitus (e.g. on insulin or an oral hypoglycemic agent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2015-04-04 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolph M. Navari, MD, PhD, FACP, Study Chair — Indiana University School of Medicine South Bend
Locations (177):
- United States (177):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Saint Mary Corwin Medical Center, Pueblo, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Sanford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital Memorial Medical Center, Daytona Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Leeward, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Waukesha Memorial Hospital, Waukesha, Illinois
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center-Sioux City, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Baptist Health Corbin, Corbin, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Botsford Hospital, Farmington, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Central Vermont Medical Center, Berlin Corners, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Cheyenne Regional Medical Center-West, Cheyenne, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Westfields Hospital/Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - William Beaumont Hospital-Royal Oak, Royal Oak, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Navari RM, Qin R, Ruddy KJ, Liu H, Powell SF, Bajaj M, Dietrich L, Biggs D, Lafky JM, Loprinzi CL. Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Jul 14;375(2):134-42. doi: 10.1056/NEJMoa1515725. PMID 27410922
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four-hundred and one (401) participants were enrolled from 46 academic or community practice institutions in the United States between August 2014 and March 2015.
Pre-assignment Details: There were eighteen participants withdrew consent (8 Olanzapine; 10 Placebo); and three participants had major violations (2 Olanzapine; 1 Placebo). All of these 21 participants were excluded from all analyses.
Groups:
- Olanzapine: Patients receive the chemotherapy drugs cisplatin or cyclophosphamide and doxorubicin as well as the following anti-nausea/vomiting drugs:
  * Ondansetron (8 mg orally or intravenously) or granisetron (1 mg intravenously or 2 mg orally) or palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (12 mg orally on the day of chemotherapy and 8 mg orally days 2, 3, 4 post chemotherapy), plus
  * Fosaprepitant (150 mg intravenously on the day of chemotherapy) or aprepitant (125 mg orally on the day of chemotherapy and 80 mg orally on days 2 and 3 post chemotherapy), plus
  * olanzapine (10 mg orally on the day of chemotherapy and 10 mg orally on days 2, 3, 4 post chemotherapy)
- Placebo: Patients receive the chemotherapy drugs cisplatin or cyclophosphamide and doxorubicin as well as usual anti-nausea/vomiting drugs:
  * Ondansetron (8 mg orally or intravenously) or granisetron (1 mg intravenously or 2 mg orally) or palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (12 mg orally on the day of chemotherapy and 8 mg orally days 2, 3, 4 post chemotherapy), plus
  * Fosaprepitant (150 mg intravenously on the day of chemotherapy) or aprepitant (125 mg orally on the day of chemotherapy and 80 mg orally on days 2 and 3 post chemotherapy), plus
  * placebo
Period: Overall Study
Arm/Group | Olanzapine | Placebo
Started | 192 | 188
Completed | 183 | 184
Not Completed | 9 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other Medical Problems | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants who started the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Placebo | Total
Number analyzed (Participants) | 192 | 188 | 380
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 86] | 56 [28 to 89] | 57 [28 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 136 | 275
  Male | 53 | 52 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 172 | 171 | 343
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 192 | 188 | 380
5-hydroxytryptamine type 3 receptor antagonist [Count of Participants; unit: Participants]
  Palonosetron | 145 | 143 | 288
  Ondansetron | 46 | 44 | 90
  Granisetron | 1 | 1 | 2
Chemotherapy regimen [Count of Participants; unit: Participants]
  Cisplatin-containing regimen | 71 | 65 | 136
  Anthracyline and cyclophosphamide | 121 | 123 | 244
Primary site of disease [Count of Participants; unit: Participants]
  Breast | 120 | 122 | 242
  Lung | 27 | 22 | 49
  Other | 45 | 44 | 89
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 149 | 144 | 293
  1=Symptomatic and fully ambulatory | 40 | 41 | 81
  2=Symptomatic, <50% in bed during the day | 2 | 3 | 5
  Not assessed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With no Nausea
Description: No nausea was defined as a response of 0 in the nausea item of Nausea and Vomiting Daily Diary/Questionnaire in the acute (0-24 hours), delayed (25-120 hours) and overall (0-120 hours) periods after chemotherapy.
Time Frame: 0 to 120 hours after chemotherapy
Population: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations and had Nausea data.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 183 | 181
percentage of participants
  0-24 hours after chemotherapy | 73.8 | 45.3
  25-120 hours after chemotherapy: number analyzed (Participants) | 177 | 177
  25-120 hours after chemotherapy | 42.4 | 25.4
  0-120 hours after chemotherapy: number analyzed (Participants) | 177 | 178
  0-120 hours after chemotherapy | 37.3 | 21.9

2. Secondary Outcome: Median Nausea Scores
Description: Nausea scores was measured using a visual-analogue scale ranging from 0 (none) to 10 (as bad as it can be).
Time Frame: Baseline and Day 2 to Day 6 after chemotherapy
Population: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations and had Nausea data at each time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 190 | 188
units on a scale
  Baseline | 0 [0 to 7] | 0 [0 to 9]
  Day 2: number analyzed (Participants) | 183 | 181
  Day 2 | 0 [0 to 10] | 1 [0 to 10]
  Day 3: number analyzed (Participants) | 182 | 180
  Day 3 | 0 [0 to 9] | 1 [0 to 10]
  Day 4: number analyzed (Participants) | 179 | 179
  Day 4 | 0 [0 to 8] | 1 [0 to 9]
  Day 5: number analyzed (Participants) | 179 | 174
  Day 5 | 0 [0 to 10] | 1 [0 to 10]
  Day 6: number analyzed (Participants) | 176 | 174
  Day 6 | 0 [0 to 9] | 1 [0 to 10]

3. Secondary Outcome: Proportion of Patients With Complete Response
Description: Complete response was defined as no emetic episodes and no use of rescue medication during the acute (0-24 hours), delayed (25-120 hours) and overall (0-120 hours) periods as measured by the Nausea and Vomiting Daily Diary/Questionnaire.
Time Frame: 0 to 120 hours after chemotherapy
Population: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations and had data on emetic and use of rescue medication questions.
Measure: Number; unit: percentage of participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 182 | 181
percentage of participants
  0-24 hours after chemotherapy | 85.7 | 64.6
  25-120 hours after chemotherapy: number analyzed (Participants) | 163 | 168
  25-120 hours after chemotherapy | 66.9 | 52.4
  0-120 hours after chemotherapy: number analyzed (Participants) | 162 | 170
  0-120 hours after chemotherapy | 63.6 | 40.6

4. Secondary Outcome: Mean Scores of Potential Toxicities Related to Olanzapine as Measured by the Nausea and Vomiting Daily Diary/Questionnaire
Description: Patients were asked to record daily levels of undesired sedation and appetite increase using a visual-analogue scale ranging from 0 (none) to 10 (as bad as it can be).
Time Frame: Baseline and day 2 to 6 days after chemotherapy
Population: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations and had toxicities data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 190 | 188
units on a scale
  Baseline Undesired Sedation | 0.4 (1.2) | 0.5 (1.5)
  Day 2 Undesired Sedation: number analyzed (Participants) | 181 | 181
  Day 2 Undesired Sedation | 2.3 (3.2) | 1.2 (2.2)
  Day 3 Undesired Sedation: number analyzed (Participants) | 182 | 180
  Day 3 Undesired Sedation | 1.6 (2.5) | 1.4 (2.3)
  Day 4 Undesired Sedation: number analyzed (Participants) | 179 | 179
  Day 4 Undesired Sedation | 1.5 (2.3) | 1.4 (2.3)
  Day 5 Undesired Sedation: number analyzed (Participants) | 179 | 173
  Day 5 Undesired Sedation | 1.2 (2.1) | 1.2 (2.1)
  Day 6 Undesired Sedation: number analyzed (Participants) | 175 | 174
  Day 6 Undesired Sedation | 0.9 (1.8) | 1.3 (2.2)
  Baseline Appetite Increase: number analyzed (Participants) | 190 | 187
  Baseline Appetite Increase | 0.6 (1.7) | 0.3 (0.9)
  Day 2 Appetite Increase: number analyzed (Participants) | 183 | 181
  Day 2 Appetite Increase | 0.7 (1.6) | 0.5 (1.5)
  Day 3 Appetite Increase: number analyzed (Participants) | 182 | 180
  Day 3 Appetite Increase | 0.7 (1.5) | 0.6 (1.7)
  Day 4 Appetite Increase: number analyzed (Participants) | 179 | 179
  Day 4 Appetite Increase | 1.0 (1.8) | 0.7 (1.7)
  Day 5 Appetite Increase: number analyzed (Participants) | 179 | 174
  Day 5 Appetite Increase | 1.0 (1.8) | 0.7 (1.7)
  Day 6 Appetite Increase: number analyzed (Participants) | 176 | 174
  Day 6 Appetite Increase | 1.1 (2.0) | 0.7 (1.7)

5. Secondary Outcome: Frequency of Rescue Medication
Description: Patients were asked to record daily number of extra nausea/vomiting pills taken because they developed nausea/vomiting in the following categories: None, One, Two, More than two in Nausea and Vomiting Daily Diary Questionnaire.
Time Frame: Day 2 to Day 6 after chemotherapy
Population: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations and had rescue medication data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Olanzapine | Placebo
Number analyzed (Participants) | 182 | 181
Participants
  Day 2: None | 156 | 117
  Day 2: Once | 21 | 35
  Day 2: Twice | 3 | 19
  Day 2: More than twice | 2 | 10
  Day 3: number analyzed (Participants) | 180 | 178
  Day 3: None | 158 | 124
  Day 3: Once | 11 | 24
  Day 3: Twice | 7 | 20
  Day 3: More than twice | 4 | 10
  Day 4: number analyzed (Participants) | 170 | 176
  Day 4: None | 141 | 124
  Day 4: Once | 16 | 24
  Day 4: Twice | 10 | 17
  Day 4: More than twice | 3 | 11
  Day 5: number analyzed (Participants) | 173 | 171
  Day 5: None | 145 | 131
  Day 5: Once | 19 | 23
  Day 5: Twice | 5 | 7
  Day 5: More than twice | 4 | 10
  Day 6: number analyzed (Participants) | 171 | 171
  Day 6: None | 143 | 130
  Day 6: Once | 12 | 16
  Day 6: Twice | 12 | 11
  Day 6: More than twice | 4 | 14

ADVERSE EVENTS:
Time Frame: Day 2 to Day 4 after chemotherapy
Description: All participants who met eligibility criteria, did not cancel prior to receiving treatment, had no major violations. Adverse events were not assessed on seven participants due to participants went off treatment on day 1 of chemotherapy (3 Olanzapine, 3 Placebo) or nurse was not able to reach one Olanzapine participant for the assessment.
Arm/Group | Olanzapine | Placebo
Serious Adverse Events (participants affected / at risk) | 3/188 | 0/185
Other Adverse Events (participants affected / at risk) | 44/188 | 36/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=188) | Placebo (N=185)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=188) | Placebo (N=185)
Palpitations (Cardiac disorders) | 0 (0) | 1 (3)
Blurred vision (Eye disorders) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 3 (4) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (8)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 9 (17)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (13) | 9 (12)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (6) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (5) | 11 (13)
Somnolence (Nervous system disorders) | 20 (29) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less